CLINICAL TRIAL: NCT04403815
Title: Determinants of Operator Radiation Exposure During Percutaneous Coronary Procedures According to Vascular Access: the RADIANT II Observational Study
Brief Title: Radiation Exposure During Coronary Procedures According to Vascular Access
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Azienda ULSS 3 Serenissima (Other)
Responsible Party: Sponsor
Other Study IDs: 1136
Record Dates: First submitted 2020-05-15; First posted 2020-05-27 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Radiation Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- right radial access: diagnostic coronary angiography and/or PCI performed through right wrist and distal ("snuffbox") radial access
  Interventions: Procedure: vascular access for coronary procedures
- left distal radial access: diagnostic coronary angiography and/or PCI performed through left distal ("snuffbox") radial access
  Interventions: Procedure: vascular access for coronary procedures

INTERVENTIONS:
Procedure: vascular access for coronary procedures — comparison of x-rays exposition of interventional cardiologist according to vascular access used

SUMMARY:
Trial's objective is to evaluate:

i. if there's any difference between the operator radiation exposure during diagnostic coronary angiography and/or percutaneous coronary intervention (PCI) performed through right-side artery accesses (wrist transradial access and distal transradial access) versus left distal radial artery access ii. the relationship between operator radiation exposure and other clinical and procedural characteristics, to assess independent predictors of operator radiation exposure. Design of the study: prospective multicenter observational cohort registry (OCR).

The purpose of this OCR is to assess the radiation exposure of interventional cardiologist during a diagnostic coronary angiography and/or PCI according to vascular access used (see above). Coronary angiography and PCI will be performed according to usual practice

DETAILED DESCRIPTION:
Patient population:

During 6 months, at least 1000 consecutive patients (age > 18 years) referred for diagnostic coronary angiography in up to 10 centers in Italy involving a minimum of 4 operators will be enrolled. To be qualified as expert, operators should have performed at least 250 transradial procedure/year in the previous 3 years and have performed at least 20 right and left distal radial procedures.

Demographic and medical history data of patients including age, sex, history of diabetes mellitus, hypertension, height and weight will be collected. Height and weight of operators will be also recorded. Type of angiographic system will be recorded. Procedural data as contrast medium amount, subclavian tortuosity, numbers of diagnostic and guiding catheters and numbers of cine-angiographic acquisitions (frames) will be also recorded.

Subclavian tortuosity will be classified as:

* Grade 1: tortuosity or calcification of the subclavian artery that can be crossed by a standard 0.035" nonhydrophilic wire facilitated with deep inspiration
* Grade 2: tortuosity or calcification of the subclavian artery that can be crossed with a 0.0035" hydrophilic wire and a standard diagnostic catheter
* Grade 3: tortuosity or calcification of the subclavian artery or congenital anomalies that require a 0.035" stiff wire and a standard catheter
* Grade 4: severe tortuosity and/or calcification of the subclavian artery or congenital anomalies preventing the catheter or guide to reach the aortic valve plane or engage the coronary ostia with a stiff wire Subclavian tortuosity > grade 2 will be considered as significative. Type of catheters and the number of views for angiography and PCI will be left to the discretion of the operator. Lead shields placed under the catheterization table, as well as ceiling mounted lead shields, will be used in every procedure. Procedural success is defined as completion of the procedure through the intended arterial access. Crossover, if needed, is permitted to femoral access or to contralateral arm or approach.

Arterial access protocol:

Right radial access: radial artery access will be obtained with a 20-gauge Teflonsheated needle using the Seldinger or the counter puncture technique. An introducer sheath is inserted in the radial artery according to local practice. An intra-arterial vasodilator cocktail will be administered consisting of ntroglycerin 200 mcg and verapamil 5 mg after sheath insertion. 5000 IU of unfractioned heparin will be administered intravenously after sheath insertion, and adequately adjusted in case of interventions. The introducer sheath will be removed at the end of the procedure, and a mechanical or inflatable pressure band will be applied to the access site to achieve hemostasis.

Distal radial accesses: following distal radial artery palpation, 1 of the 2 possible puncture sites (anatomic snuffbox or in the first intermetacarpal space) is chosen. In case of left-side access, the left hand is bent toward the left groin with support below the left elbow to ensure patient's comfort. The operator is positioned at the right side of the patient. To favor a shift of the distal radial artery to the surface of the fossa, the patient is asked to grasp his or her thumb under the other 4 fingers or to hold a roll of gauze, a 20 ml syringe, or the handle of a dedicated system. After disinfection and local anesthesia, the artery is punctured according to operator preference and/or experience using a micropuncture needle or a cannula-over-needle. An introducer sheath (preferably a slender introducer sheath) is inserted in the radial artery according to local practice. An intra-arterial vasodilator cocktail will be administered consisting of nitroglycerin 200 mcg and verapamil 5 mg after sheath insertion. 5000 IU of unfractioned heparin will be administered intravenously after sheath insertion, and adequately adjusted in case of interventions.

Coronary catheterization:

Angiographic systems were set according to the standard of the operators, and the field of view or fluoroscopic and cine-acquisition speed will be recorded for each procedure. The diagnostic procedures will be performed using a standard sequence of 3 projections for the right coronary artery and maximum 6 projections for the left coronary artery. Differently, the percutaneous coronary interventions will be performed according to the lesion and to the operator preference.

Vascular access as well as the sheath selection, catheter curve used, and the use of adjunctive tools will be at the discretion of the operator involved in the procedure.

In all procedures, standard operator radioprotection will be ensured using a lead apron, a thyroid lead collar, lower body x-ray curtain fixed on the angiographic table, an upper mobile leaded glass suspended from the ceiling, and leaded glasses. The use of adjunctive protective drapes to reduce operator radiation exposition ws left to the operator's discretion

Radiation measurement:

Radiation measures collected are fluoroscopy time (expressed in minutes), the AK (expressed in mGy) and the DAP (expressed in Gy*cm2). The number of acquired cineangiograms will be recorded. Fluoroscopy and cineangiography will be performed at 7.5 or 15 frames/s according to operators' preferences.

Operator radiation exposure is measured for each participating operator using 1 dedicated electronic dosimeter (PM1610B; Polimaster, Vienna, Austria) to be worn at mid-thorax level, in the breast pocket outside the lead apron, and expressed in µSy. The radiation and operator measures will be recorded at the beginning and the end of each procedure. For those patients who undergo a PCI after the diagnostic procedure, the measures of fluoroscopy time, DAP, and dose of the wearable dosimeters will be reset after the end of the diagnostic procedure and restart at the beginning of the PCI. To take into account possible differences in patient radiation dose affecting the operator exposure, the DAP-normalized operator dose will be also calculated.

The equivalent dose at the thorax will be also converted in operator effective dose dividing it by a factor of 33 according to apron thickness, 0.5 lead equivalent with a tube voltage under the table. Patient effective dose will be calculated using a conversion factor of 0.20 mSv/Gy*cm2.

Statistical Hypothesis and analysis:

the null hypothesis is that ld-TRA exposure to radiation is the same as right-side TRA (access site at the wrist and at the anatomical snuffbox of the right hand). In the previous RADIANT study right-side TRA was associated with a mean operator exposition of 13 µSy (SD +10 µSy); hence, to detect non-inferiority between the two groups (risk of type I error 5%, risk of type II error 80%, non-inferiority limit 3 µSy) at least 138 per group are needed. The alternative hypothesis is that ld-TRA exposure is reduced compared to rightside TRA. The amount of this reduction is to be determined. An arbitrary period of 6 months should be sufficient to record the radiological exposition in at least 1000 procedures. Taking into account possible crossover between groups, a minimum proportion of 20% of procedures through distal left radial artery PCIs was mandated to guarantee adequate numerosity of the group. Kolmogorov-Smirnov analysis will be performed to evaluate the distribution of each variable analyzed. Categorical variables will be analyzed using chi-square test, and continuous variables will be analyzed using analysis of variance for normally distributed variables and Kruskal-Wallis test for variables with distribution that were not normal. If needed, log-transformation of non-normal variables will be performed. Hierarchical linear regression will be used to identify independent predictors of radiation exposure, entering control variables found to be significantly associated with radiation exposure on univariate analysis. Propensity score matching will be performed to minimize the risks of imbalances due to variation in the complexity of the diagnostic or therapeutic procedures within each operators. Prespecified analysis of subgroups (diagnostic coronary angiography vs PCI, expert operators vs fellows, use of adjunctive drapes, physical characteristics of operators) could be planned.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted for coronary diagnostic angiography in the setting of valvular disease, stable angina, suspected coronary artery disease, acute coronary syndrome with or without ST segment elevation myocardial infarction who underwent diagnostic coronary angiography through right radial, right distal radial and left distal radial access.
* patients admitted for ad-Hoc PCI through any radial access
* patients age > 18 years-old
* signed informed consent

Exclusion Criteria:

* hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all-comers undergoing to diagnostic coronary angiography and/or PCI through transradial access
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
mean operator radiation dose | 1 year
  mean operator radiation dose at the torax (expressed in µSy)

SECONDARY OUTCOMES:
patient radiation exposure | from beginning to end of coronary procedure
  Patient effective dose: operator effective dose divided by a conversion factor of 0.20 mSv/Gy*cm2
mean fluoroscopy time | 1 year
  mean fluoroscopy time (minutes)
mean DAP-normalized operator dose | 1 year
  operator radiation dose divided by DAP values
mean operator effective dose | 1 year
  Operator effective dose: operator radiation exposure divided by 0.33

IPD SHARING:
Plan to Share IPD: No